## Combining Treatment Components in Transdiagnostic Therapy for Anxiety and Depression: A Randomized Controlled Trial

Date: November 20, 2025

## Clinically meaningful improvement and deterioration

We will evaluate clinically meaningful changes in primary outcomes in two different ways. First, using a Cohen's d of 0.5 (often used as a measure of clinically meaningful change; Norman et al., 2003), and second, by calculating the Reliable Change Index (Jacobson & Truax, 1991). We will use these thresholds to determine the proportion of participants who experience a clinically meaningful improvement or deterioration (i) after receiving one treatment component and (ii) after receiving both treatment components.

## References

- Jacobson, N. S., & Truax, P. (1991). Clinical significance: A statistical approach to defining meaningful change in psychotherapy research. *Journal of Consulting and Clinical Psychology*, 59(1), 12-19. <a href="https://doi.org/10.1037/0022-006X.59.1.12">https://doi.org/10.1037/0022-006X.59.1.12</a>
- Norman, G. R., Sloan, J. A., & Wyrwich, K. W. (2003). Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. *Med Care*, 41(5), 582-592. https://doi.org/10.1097/01.Mlr.0000062554.74615.4c